CLINICAL TRIAL: NCT01107106
Title: Prospective Observational Single Arm Open-Label Multicenter Study to Assess the Safety, Tolerability and Efficacy of ellaOne® (Ulipristal Acetate) for Emergency Contraception in Postmenarcheal Adolescent Girls and Adult Women
Brief Title: Safety, Tolerability, and Efficacy of ellaOne® (Ulipristal Acetate) for Emergency Contraception in Postmenarcheal Adolescent Girls and Women
Status: Completed | Type: Observational
Sponsor: HRA Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: 2914-010; 2009-017771-21 (EudraCT Number)
Record Dates: First submitted 2010-04-12; First posted 2010-04-20 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: Contraception
Keywords: Contraceptive Methods; Female Contraception
MeSH Terms: interventions — ulipristal acetate

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adolescents: 250 postmenarcheal adolescent girls
  Interventions: Drug: ellaOne® (ulipristal acetate)
- Adults: 250 adult women
  Interventions: Drug: ellaOne® (ulipristal acetate)

INTERVENTIONS:
Drug: ellaOne® (ulipristal acetate) — one single oral dose (30 mg tablet)
  Other Names: ellaOne®
  Groups: Adolescents
Drug: ellaOne® (ulipristal acetate) — one single oral dose (30 mg tablet)
  Other Names: ellaOne®
  Groups: Adults

SUMMARY:
The purpose of this observational study is to assess the safety and tolerability of ellaOne® in routine conditions of use for emergency contraception in postmenarcheal adolescents and adult women who want to prevent pregnancy up to 5 days after unprotected sexual intercourse.

ELIGIBILITY:
Inclusion Criteria:

* Having received ellaOne® as emergency contraception at the clinical site
* Postmenarcheal adolescents or adult women
* Willing to provide information on bleeding, sexual intercourses, method of contraception, concomitant medications and adverse events for the next two menstrual periods and to complete the diary accordingly
* Willing to provide information on pregnancy outcome / delivery and newborn's health at delivery
* Able to provide written informed consent
* Willing to not participate in a clinical trial before the end of study participation

Exclusion Criteria:

* Currently participating in any interventional clinical trial (testing an Investigational Medicinal Product)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adolescents and adult women seeking emergency contraception in family planning centers and youth clinics in Sweden
Sampling Method: Non-Probability Sample
Enrollment: 579 (Actual)
Dates: Start 2010-05; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events after ellaOne® intake in routine conditions of use for emergency contraception | Two months (i.e. all along 2 menstrual cycles following ellaOne® intake)
  Collection of adverse events, concomitant treatments, length of menstrual cycle, and vaginal bleeding/spotting through follow-up contacts and a diary completed by the patient

SECONDARY OUTCOMES:
Pregnancy rate observed after taking ellaOne® in routine conditions of use for emergency contraception | Two months (i.e. during two menstrual cycles following ellaOne® intake)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - PPRM Central clinic, Denver, Colorado
  - PPRM Southwest clinic, Lakewood, Colorado
  - Elizabeth Blackwell Health Center, Philadelphia, Pennsylvania
  - Locust Health Center, Philadelphia, Pennsylvania
- Dept of Women & Child Health - Karolinska University Hospital, Stockholm, Sweden
- Brook clinic, Belfast, United Kingdom